CLINICAL TRIAL: NCT05783141
Title: Double-blind, Randomized Placebo-controlled Trial Investigating Cumulative or Even Synergistic Effects of a Novel Prebiotic Combination in Healthy Toddlers
Brief Title: Prebiotic Effects in Healthy Toddlers
Acronym: PrebiKidz
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Collaborators: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22006n-mpz
Record Dates: First submitted 2023-02-21; First posted 2023-03-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Child Development; Diet, Healthy
Keywords: Microbiota; Prebiota; Child´s health
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental formula group (Experimental): Follow-on formula supplemented with a novel prebiotic combination
  Interventions: Dietary Supplement: New prebiotic follow-on formula, randomly assigned to healthy toddlers
- Control formula group (Placebo Comparator): Follow-on formula not supplemented
  Interventions: Dietary Supplement: Standard follow-on formula, randomly assigned to healthy toddlers

INTERVENTIONS:
Dietary Supplement: New prebiotic follow-on formula, randomly assigned to healthy toddlers — Standard follow-on formula administered orally
  Other Names: supplemented with prebiotics
  Arms: Experimental formula group
Dietary Supplement: Standard follow-on formula, randomly assigned to healthy toddlers — Standard follow-on formula administered orally
  Other Names: not supplemented with prebiotics
  Arms: Control formula group

SUMMARY:
The aim of this study is to demonstrate that a dietary supplementation with a novel prebiotic combination is safe, well tolerated and able to improve overall health of toddlers.

DETAILED DESCRIPTION:
The fermentation of a novel prebiotic combination leads to a modulation of the gut microbiota composition, in particular to a growth stimulation of bifidobacteria, and the production of organic acids like lactate and short-chain fatty acids (SCFA).The efficacy of the prebiotic combination to improve toddler's digestive function will be addressed. The overall health will be assessed as a measure of reduced number of febrile days resulting in less days of absenteeism from daycare centers.

ELIGIBILITY:
Inclusion Criteria:

1. Child is healthy at the time of pre-examination
2. Child is aged between 10-36 months and attends a day care center for the duration of the intervention
3. Child attends a daycare center at the time of pre examination for at least 50%.
4. Child presents a normal defecation characteristic (according to Brussels Infant and Toddler Stool scale)
5. Weight for height z-score >-2 and <2 SD based on Flemish growth charts
6. Child and legal guardian are able and willing to follow the study instructions
7. Child is suitable for participation in the study according to the investigator/ study personnel
8. Informed written consent given by parent / legal guardian

Exclusion Criteria:

1. No legal guardian's command of any local language
2. Child with any chronic disorder or disease, e.g., defecation disorders (incl. Hirschsprung and celiac disease) metabolic or renal abnormalities as well as mental or psychomotor retardation (incl. child´s mental delay and hypotonia)
3. Child is suffering from congenital or acquired immunodeficiency
4. Food allergies or intolerances
5. Child is currently breast-fed more than once daily
6. Use of drugs (e.g. antibiotics) influencing gastrointestinal function (6 weeks before intervention)
7. Use of laxatives (4 weeks before intervention) as well as probiotic and prebiotic food supplements. Follow-on formula with L. Reuteri and/or GOS/FOS/HMO is allowed.
8. Child is suffering from an infection at the time of pre examination or previous 7 days
9. Child is currently involved or will be involved in another clinical or food study
10. Child is not suitable for participation in the study according to the study personnel´s opinion

Ages: 10 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 342 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Fever | Data collected continuously from enrollment until end of intervention (up to 90 days).
  Number of febrile days (peak temperature of forehead at least 38.0°C)
Absenteeism | Data collected continuously from enrollment until end of intervention (up to 90 days).
  Number of days of child´s absence from day care center due to infectious episodes or antibiotic treatment.

SECONDARY OUTCOMES:
Beneficial colonization | Stool sample collected at baseline and after 90 days intervention period
  Changes in fecal microbiota by 16S rRNA Sequencing
Stool consistency | Data collected continuously from enrollment until end of intervention (up to 90 days).
  Hard, formed, soft and watery stools will be assessed by the parents and day care centers in a continuous daily bowel diary using the Brussels Infant and Toddler Stool Scale
Stool frequency | Data collected continuously from enrollment until end of intervention (up to 90 days).
  Number of defecations will be assessed by the parents and day care centers in a continuous daily bowel diary using the Brussels Infant and Toddler Stool Scale
Caretaker´s absenteeism from work | Data collected continuously from enrollment until end of intervention (up to 90 days).
  Number of work days missed by the parents

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Vandenplas, Prof., Principal Investigator — Universitair Ziekenhuis Brussel; Koen Huysentruyt, Prof., Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium